CLINICAL TRIAL: NCT01226277
Title: An Open-Label, Phase I, Dose-Escalation Study Evaluating the Safety, Tolerability and Pharmacokinetics of GDC-0917 Administered Daily in Patients With Refractory Solid Tumors or Lymphoma
Brief Title: A Study Evaluating the Safety, Tolerability and Pharmacokinetics of GDC-0917 Administered to Patients With Refractory Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4914g; GO01306 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2010-10-20; First posted 2010-10-22 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Solid Cancers

ARMS (1):
- A (Experimental)
  Interventions: Drug: GDC-0917

INTERVENTIONS:
Drug: GDC-0917 — Oral repeating dose

SUMMARY:
This is an open-label, multicenter, Phase I dose-escalation study designed to assess the safety, tolerability, and pharmacokinetics (PK) of GDC-0917 in patients with refractory solid tumors or lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented, locally advanced or metastatic solid tumors or lymphoma for which standard therapy either does not exist or has proven ineffective or intolerable
* Life expectancy >/= 12 weeks
* Adequate hematologic and end organ function
* For female patients of childbearing potential and male patients with partners of childbearing potential, agreement (by patient and/or partner) to use an effective form of contraception and to continue its use for the duration of the study.

Exclusion Criteria:

* Clinically significant history of chronic liver disease, active hepatic infection, evidence of hepatic cirrhosis or Grade >/= 2 liver dysfunction not due to hepatic metastases of cancer, current alcohol abuse, active infections with hepatitis B virus, or hepatitis C virus
* Grade >/= 2 fever or associated constitutional symptoms, or a clinically significant systemic infection within the last month
* Autoimmune disease
* History of clinically significant pulmonary disease
* Need for chronic and continuous systemic or topical corticosteroids or immunosuppressive therapy within 2 weeks prior to study entry or anticipated need of continuous systemic corticosteroids or immunosuppressive therapy during study participation.
* Allergy or hypersensitivity to components of the GDC-0917 formulation
* Palliative radiotherapy within 2 weeks prior to first dose of study drug treatment in Cycle 1
* Experimental therapy within 4 weeks prior to first dose of study drug treatment in Cycle 1
* Major surgical procedure or significant traumatic injury within 4 weeks prior to first dose of study drug treatment in Cycle 1, or anticipation of the need for major surgery during the course of study treatment
* Prior anti-cancer therapy within 4 weeks before the first dose of study drug treatment in Cycle 1
* All acute drug-related toxicities must have resolved prior to study entry, except for alopecia and Grade 1 neuropathy
* Current severe, uncontrolled systemic disease excluding cancer
* History of clinically significant cardiac dysfunction
* History of malabsorption or other condition that would interfere with enteral absorption
* Any history of active GI bleeding within the past 6 months prior to screening
* Known HIV infection
* Uncontrolled ascites, due to diseases other than cancer, requiring weekly large-volume paracentesis for 3 consecutive weeks prior to enrollment
* Pregnancy, lactation, breastfeeding or unwillingness to use birth control during the study and for 3 months after the last dose of GDC-0917
* Known brain metastases that are untreated, symptomatic, or require therapy to control symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Changes in vital signs, ECGs, and clinical laboratory results | Throughout study or until early discontinuation
Incidence and nature of dose-limiting toxicities and adverse events of special interest | Throughout study or until early discontinuation
Incidence, nature, and severity of all adverse events and serious adverse events | Throughout study or until early discontinuation

SECONDARY OUTCOMES:
Pharmacokinetic parameters of GDC-0917 (including total exposure, maximum and minimum serum concentration, time to maximum observed plasma concentration, elimination of half-life, accumulation at steady-state) | Throughout study or until early discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Chia Portera, M.D., Ph.D., Study Director — Genentech, Inc.
Locations (2):
- United States (2):
  - Nashville, Tennessee
  - San Antonio, Texas